CLINICAL TRIAL: NCT05474183
Title: The Role of Ketamine and Dexmedetomidine in Opioid-Sparing Analgesia and Sedation in Adult Patients After Cardiac Surgery. A Randomized Clinical Trial
Brief Title: The Role of Ketamine and Dexmedetomidine in Opioid-Sparing Analgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fayoum University Hospital (Other)
Responsible Party: Principal Investigator, Mohamed Ahmed Hamed, ASSOCIATE PROFESSOR OF ANESTHESIA, Fayoum University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H123
Record Dates: First submitted 2022-06-29; First posted 2022-07-26 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Ketamine-Induced Mood Disorder
Keywords: ketamine; dexmedetomidine; Analgesia; Cardiac Surgery; Sedation
MeSH Terms: conditions — Agnosia | interventions — Ketamine; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group (K) (Active Comparator): Group (K): (n=30) will receive ketamine infusion 1-2 μg/kg/min (0.12 mg/kg/h) titrated to desired level of sedation.
  Interventions: Drug: Ketamine
- Group (D) (Active Comparator): Group (D): (n=30) will receive Dexmedetomidine infusion 0.1- 0.2 μg/kg/hour titrated to desired level of sedation.
  Interventions: Drug: Ketamine
- Group (C) (Placebo Comparator): Group (C): (n=30) will receive fentanyl only.
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — drug
  Other Names: dexmedetomidine

SUMMARY:
Optimal multimodal opioid-sparing analgesic technique is considered as one of the most important Enhanced recovery pathways (ERPs) or enhanced recovery after surgery (ERAS) interventions that mitigate the undesirable effects of surgical stress response. Implementation of ERP has been shown to reduce postoperative complications and shorten the hospital LOS.

DETAILED DESCRIPTION:
In this study, the investigator hypothesizes that by using continuous infusion of ketamine or dexmedetomidine in addition to NSAIDs, the investigator can reduce or completely eliminate opioid use in adult patients after cardiac surgery.

The anesthesia technique was composed of the following 10 steps:

1. Premedication with oral Pregabalin 75 mg the night before surgery;
2. For induction and maintenance of anesthesia: - Midazolam 0.02- 0.05 mg/kg bolus, -Fentanyl (cumulative dose 5-15 μg/kg), followed by continuousInfusion of Fentanyl; 2-3 μg/kg /h as a maintenance dose, Rocuronium: (0.6-1.0 mg/kg - intubation dose, followed by continuous Infusion of Rocuronium; 0.075-0.15 mg/kg/h as a maintenance dose, and Sevoflurane in a dose of 0.8-1.0 (MAC).
3. Ventilation: Lung protective ventilation (Vt 6 ml/kg predicted body weight, + PEEP 5, + FiO2 60%), and we conducted a recruitment maneuver in order to prevent atelectasis.
4. Monitoring: Routine monitors (ECG, SpO2, arterial line inserted using local anesthesia for pressure monitor and repeated ABG, Central line inserted after induction of anesthesia for monitoring CVP, ETCO2, core temperature through urinary catheter, and Activated Clotting Time (ACT) for monitoring of coagulation). Cerebral oximetry, and Bispectral Index (BIS) as an indicator of depth anesthesia was kept between 40 and 60. (5) Cardiopulmonary Bypass (CPB): Goal directed perfusion maintaining MAP ≥ 60, using Phenylephrine and Norepinephrine infusion. Additional propofol infusion (25 - 50µg/kg/min) was administered during CPB to maintain BIS between 40 and 60. Smooth conduct of CPB, with Mild hypothermia (28°C 32°C). Rewarming at the end of the procedure, Goal postop temperature >36 °C.

(6) Perioperative Glycemic Control: Insulin infusion, and the perioperative Goal glucose ≤ 150 - 180.

(7)Perioperative hemoglobin concentration: Goal hemoglobin transfusion trigger: 7.5 regardless of patient Age and Comorbidity. (8) Protamine: Post CPB protamine (heparin reversal) given up to the full dose (5 mg/kg after test dose) to return to baseline ACT.

(9) Multimodal analgesia: In addition to continuous infusion of Fentanyl, at the end of the surgery, Paracetamol: 1 gm IV infusion over 15 min was administered with the sternum closure, and Surgical Incision Field Block using 30 ml of Bupivacaine 0.5% just before dressing. The patient will then be transferred intubated to Surgical ICU (SICU). (10) In SICU: Postoperative analgesia will be carried out for all groups. All patients will receive IV fentanyl via patient-controlled analgesia (PCA) with (10 µg.mL-1, with a bolus of 15 µg, and lockout 10 minutes, maximum cumulative dose of 90µ.hr-1 and no background dose). Before extubation, analgesia will be given as nurse-controlled analgesia (NCA) with the same regimen, depending on the sudden rise in HR or MABP ≥20% of the baseline. The total of 24 h. opioid consumption will be recorded.

At this step, and for opioid-sparing analgesia and sedation, using the sealed envelope technique, patients will be randomly divided into three groups: Group (K): (n=30) will receive ketamine infusion of 1-2 μg/kg/min (0.12 mg/kg/h) titrated to the desired level of sedation. Group (D): (n=30) will receive Dexmedetomidine infusion 0.1- 0.2 μg/kg/hour titrated to desired level of sedation. Group (C): (n=30) will receive fentanyl only. All hemodynamic monitors used intraoperatively are continued in SICU, and in addition, the following parameters are used to monitor the level of analgesia and sedation -During mechanical ventilation: Richmond Agitation-Sedation Scale

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 65 years
* Ejection fraction (EF) > 35%
* Elective isolated CABG
* Valve surgery, Atrial septal defect (ASD) closure
* Cross clamp time ≤ 90 min
* Cardiopulmonary bypass time ≤ 120 min.

Exclusion Criteria:

* Poor left ventricular function with intra-aortic balloon pump support
* Recent myocardial infarction (last seven days)
* Combined procedure (i.e., CABG + other heart/vascular procedure)
* Emergency surgery, and Redo surgery,Hepatic or renal failure, creatinine >1.5 -History of neurological disorders or convulsions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-08-05 (Actual); Primary Completion 2023-05-10 (Actual); Study Completion 2023-05-20 (Actual)

PRIMARY OUTCOMES:
The total postoperative fentanyl consumption (μg) | the first 48 hours postoperative
  the total doses of postoperative fentanyl consumption in (μg)

SECONDARY OUTCOMES:
Duration of mechanical ventilation | the first 48 hours postoperative
  Duration of mechanical ventilation (day)

CONTACTS AND LOCATIONS:
Locations (1):
- Fayoum University hospital, Al Fayyum, Faiyum Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
no plane

REFERENCES:
- [Background] Gan TJ. Poorly controlled postoperative pain: prevalence, consequences, and prevention. J Pain Res. 2017 Sep 25;10:2287-2298. doi: 10.2147/JPR.S144066. eCollection 2017. PMID 29026331
- [Background] Chapman CR, Vierck CJ. The Transition of Acute Postoperative Pain to Chronic Pain: An Integrative Overview of Research on Mechanisms. J Pain. 2017 Apr;18(4):359.e1-359.e38. doi: 10.1016/j.jpain.2016.11.004. Epub 2016 Nov 28. PMID 27908839